CLINICAL TRIAL: NCT04964323
Title: Pyruvate Kinase Deficiency Global Longitudinal Registry: Patient-Reported Outcomes
Brief Title: Pyruvate Kinase (PK) Deficiency Global Longitudinal Registry: Patient-Reported Outcomes (PRO)
Acronym: PKD
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment and participant compliance with surveys.
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG348-C-015
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pyruvate Kinase Deficiency; Pyruvate Kinase Deficiency Anemia; Anemia; Anemia, Hemolytic
Keywords: Glycolytic enzymopathy; Congenital Nonspherocytic Hemolytic Anemia; PKD; CNSHA
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia; Anemia, Hemolytic; Anemia, Hemolytic, Congenital Nonspherocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 96 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PK Deficiency Diagnosed: Participants previously diagnosed with PK deficiency in Study AG348-C-008 (NCT03481738), will receive routine clinical care.

SUMMARY:
The primary objective of this study is to understand and characterize the health-related quality of life (HRQoL) and disease burden of adult participants with PK deficiency receiving routine clinical care. This study is an observational (i.e., noninterventional), longitudinal, multicenter, global registry for participants with PK deficiency, a rare nonspherocytic hemolytic anemia.

This study will be open for enrollment for 2 years and all enrolled participants will be followed prospectively for up to 96 weeks.

Data will be collected from participants who have provided informed consent and authorization pursuant to applicable laws and regulations.

DETAILED DESCRIPTION:
Participants aged ≥18 years and previously enrolled in Study AG348-C-008 (NCT03481738) will be eligible to participate in this study. Data will be submitted via electronic patient-reported outcomes (ePRO) application.

All data collection efforts will abide by this protocol and be prospectively disclosed in the study informed consent. This study, with the appropriate participant (and or parent/guardian) consent/assent, may incorporate retrospective data from other properly consented studies done for the purpose of examining the longitudinal natural history of PK deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to (≥)18 years of age;
* Participant must be enrolled in Study AG348-C-008.

Exclusion Criteria:

- Participant is enrolled in an Agios-sponsored clinical study involving treatment with a pyruvate kinase activator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at multiple sites in North America and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pyruvate Kinase Deficiency Diary (PKDD) Score | Baseline, up to Day 672
  The PKDD is a 7-item measure of the core signs and symptoms of PK deficiency. The score range is 25 to 76, with higher scores indicating a higher disease burden.
Change from Baseline in Pyruvate Kinase Deficiency Impact Assessment (PKDIA) Score | Baseline, up to Day 672
  The PKDIA is a 12-item measure of the impacts of PK deficiency on patients' HRQoL. The score range is 30 to 76, with higher scores indicating a higher disease burden.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI: SHP) 2.0 Score | Baseline, up to Day 672
  WPAI:SHP is a 6-question participant-rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss, and daily activity impairment attributable to PK deficiency for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Change from Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) | Baseline, up to Day 672
  FACT-An is composed of five subscales: Physical Well-Being [score range 0-28], Social/Family Well-Being [score range 0-28], Emotional Well-Being [score range 0-24], and Functional Well-Being [score range 0-28] and specific questions concerning anemia [score range 0-80]. The score at each item is summed. The sum is multiplied by the number of items in the subscale and then divided by the number of items answered. This produces the subscale score. The subscale scores are added to derive a total score [score range 0-188]. A higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (5):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Infantil Universitario Niño Jesus - PIN, Madrid, Spain
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No